CLINICAL TRIAL: NCT06278259
Title: Telerehabilitation Program Bases Aerobic and Baduanjin Exercises on Cognition , Sleep Quality and Physical Performance in Post Stroke Elderly Patients
Brief Title: Telerehabilitation Program Bases Aerobic and Baduanjin Exercises in Post Stroke Elderly Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, marwa mahmoud elsayed mahmoud, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005023
Record Dates: First submitted 2024-02-14; First posted 2024-02-26 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The telerehabilitation program is moderately intense aerobic exercise 3 times per week and included 3 parts: warm-up, central part, and cool-down. Each session : 30 min, 3 sessions/ week for 3 months.With the Baduanjin exercise program is delivered individually, at each patient's home, through telerehabilitation, with direct remote supervision by a physiotherapist
  Interventions: Other: Telerehabilitation program bases aerobic and Baduanjin exercises
- control group (Active Comparator): The control group will receive the same aerobic exercises only
  Interventions: Other: Telerehabilitation program bases aerobic exercises

INTERVENTIONS:
Other: Telerehabilitation program bases aerobic and Baduanjin exercises — It is an interventional study in which 68 stroke patients are estimated to enroll according to random allocation and divided into two groups. The study group participants involve in Telerehabilitation sessions is based on aerobic exercises, guided by video. The telerehabilitation program is aerobic exercise 3 times per week for 3 months. With the Baduanjin exercise program is delivered individually, at each patient's home, through telerehabilitation, with direct remote supervision by a physiotherapist
  Arms: experimental group
Other: Telerehabilitation program bases aerobic exercises — The telerehabilitation program is aerobic exercise 3 times per week for 3 months.
  Arms: control group

SUMMARY:
It is an interventional study in which 68 stroke patients are estimated to be enrolled according to random allocation and will be divided into two groups. The study group participants will be involved in Telerehabilitation sessions, which will be based on aerobic exercises, guided by video with the Baduanjin exercise program; the control group will receive the same aerobic exercises only

DETAILED DESCRIPTION:
It is an interventional study in which 68 stroke patients are estimated to enroll according to random allocation and will be divided into two groups. The study group participants will be involved in telerehabilitation sessions based on aerobic exercises guided by video. The telerehabilitation program will be moderately intense aerobic exercise 3 times per week and will be 3 sessions/week for 3 months.

. The exercise intensity of each telerehabilitation session will be individually adjusted by the participants' Modified Borg perceived exertion and maximum heart rate. The Baduanjin exercise program is delivered individually, at each patient's home, through telerehabilitation, with direct remote supervision by a physiotherapist. The control group will receive the same aerobic exercises only.

ELIGIBILITY:
Inclusion Criteria:

* • The subject selection will be according to the following criteria:

  * All Patients of this study will be diagnosed as stroke and the diagnosis will be confirmed by computed tomography or MRI (El-Tamawy et al., 2021).
  * Age of patients will be more than or equal 65years (males and females).
  * All patients will be hemodynamically stable.

Exclusion Criteria:

* • The potential participants will be excluded if they meet one of the following criteria:

  * Patients who cannot follow instructions as sensory aphasia, blindness, dementia, and deafness.
  * Patients with any orthopedic, neurological, or chest disorders that affect trunk muscles control or cause respiratory disorders as COPD.
  * Patients with psychiatric disorders.
  * Patients with unstable cardiovascular conditions.
  * uncontrolled hypertension, or other concomitant respiratory diseases
  * participate at any research or rehabilitation program during the period of this study

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-11-28 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
six-minute walk test | 12 weeks
  The 6MWT is a reliable and good measure of functional capacity. The test will be carried out according to the guidelines set forth by the American Thoracic Society (ATS).

SECONDARY OUTCOMES:
Cognitive function | 12 weeks
  mini mental state examination
sleep quality | 12 weeks
  The Pittsburgh Sleep Quality Index
functional independence measure | 12 weeks
  FIM was developed to measure the ability of stroke patients to do daily tasks to assess changes in their functional status. The 18 items consist of 13 items that define a motor ability disorder
physical function | 12 weeks
  physical performance battery
berg balance scale | 12 weeks
  A common, standardized tool for assessing balance in stroke patients is the BBS. The scale has 14 components, including transfers, standing on one leg, standing to sitting, standing without assistance, and sitting to standing.

CONTACTS AND LOCATIONS:
Overall Officials: marwa elsayed, PhD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Yes
sharing
Supporting Information: Study Protocol
Time Frame: one year
Access Criteria: after acceptance of the publishing journal
URL: https://www.ekb.com